CLINICAL TRIAL: NCT03550495
Title: A Multidisciplinary Delirium Prevention Strategy Involving Psychiatry in the Intensive Care Unit (ICU): Effects on Delirium Incidence and Outcomes
Brief Title: A Multidisciplinary Delirium Prevention Strategy Involving Psychiatry in the ICU
Acronym: ICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Catherine Kuza, Clinical Assistant Professor, University of Southern California
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HS-17-00617
Record Dates: First submitted 2018-05-02; First posted 2018-06-08 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Delirium
Keywords: ICU delirium; prevention; psychiatry
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Intervention Model Description: This is a prospective, single institution, controlled, pilot study of patients admitted to the 7W ICU which will compare the incidence and delirium rates among patients undergoing routine care before intervention (no routine psychiatric involvement) (control group) and patients after the intervention (psychiatry team rounding with the ICU team daily) (intervention group) . Randomization is not possible for this study; although block randomization was considered, it will result in sub-optimal data subject to bias.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Patients will undergo standard of care including the use of the ABCDEF bundle; psychiatry team will not be involved on daily ICU rounds.
- Intervention (Experimental): Patients will receive standard ICU care, including the use of the ABCDEF bundle, but will also receive the intervention of psychiatry involvement; the psychiatry team will participate in daily ICU rounds with the ICU team to help identify, prevent, and treat ICU delirium and identify other psychiatric disorders which may be otherwise undetected by the ICU team.
  Interventions: Behavioral: psychiatry involvement

INTERVENTIONS:
Behavioral: psychiatry involvement — See arm description.
  Arms: Intervention

SUMMARY:
Delirium affects up to 80% of intensive care unit (ICU) patients and is associated with longer hospital stays, increased morbidity and mortality, and increased costs. There is no FDA-approved treatment for delirium; the most effective strategy is prevention by nonpharmacological methods. The investigators propose to study a comprehensive delirium prevention bundle that has been effective against delirium in preliminary studies in elderly in-hospital patients and elderly ICU patients. This delirium prevention bundle includes the novel addition of psychiatrists to daily ICU rounds, as these professionals are specially trained to screen for latent mental illness and provide treatment for these illnesses. The effects of daily psychiatric evaluation of ICU patients has never been systematically studied, as ICU professionals are well-equipped to manage ICU delirium. Psychiatric consultation is reserved for severe and/or refractory cases of delirium. The investigators hypothesize that a multidisciplinary rounding approach including psychiatry within the ICU team will help diagnose psychiatric components that may contribute to delirium at an earlier time point, and thus can reduce the incidence and duration of delirium. The investigators also hypothesize that the proposed multidisciplinary approach will shorten hospital and ICU lengths of stay, duration of mechanical ventilation, and decrease in-hospital mortality.

DETAILED DESCRIPTION:
This is a prospective, single institution, controlled pilot study of adult patients admitted to the surgical ICU. A sample size of 104 (52 per group) is targeted. Patients in the control group will undergo usual care which includes ABCDEF bundle (Appendix 1) use, including daily delirium screening using the CAM-ICU score (Appendix 2), but will not have routine psychiatric involvement. Patients in the intervention group will also have ABCDEF bundle performed, and additionally have psychiatry routinely participating in ICU rounds. A member of the psychiatry team (attending, resident, or fellow) will round with the surgical ICU team in the surgical ICU daily. On a daily basis, the ICU attending will review the list of the ICU patients with the psychiatry team to determine if there are any changes to the patient's management required.

Inclusion criteria are: 1. any patient >18 years of age admitted to the surgical ICU for >48 hours; 2. Patients admitted to the ICU <24 hours who have been in the hospital >48 hours; 3. Patients who return to the ICU after being discharged from the ICU to the floor due a complication or need for higher acuity care. Exclusion criteria are: 1. Patients in whom CAM-ICU cannot be performed (severe dementia, stroke or other neurological condition, encephalopathy, mental retardation, severe psychiatric disorder, vegetative state, severe traumatic brain injury, deaf/blind, etc.); 2. Vulnerable patient populations (i.e. transplant recipients); 3. Patients who don't speak or understand English; 4. Current alcohol or substance abuse. Patients will be screened for eligibility on rounds daily. Study personnel will obtain informed written consent from patients or their families.

A psychiatry attending, psychiatry resident, or psychiatry nurse practitioner will round with the surgical ICU team on 7W daily until the target subject enrollment # of 52 is achieved. On a daily basis, the ICU attending will review the list of the ICU patients with the psychiatry team to determine if there are any changes to the patient's management required. The ABCDEF bundle will be implemented on daily rounds, which includes daily screening for delirium using the CAM-ICU scale.

Data which will be collected includes: age, gender, body mass index, history or alcohol or substance abuse, admitting diagnosis, dementia, comorbid conditions, admitting SOFA score, deliriogenic medications used during study enrollment, the interventions/medications used to treat delirium as designated by psychiatry (in intervention group) and the ICU team (control group), and the number of days from admission to study enrollment. Data on the incidence of ICU delirium, duration of delirium/mechanical ventilation, in-house mortality, ICU and total hospital length of stay will also be collected.

Descriptive statistics, including Student's t-test or Mann-Whitney U-test, for continuous variables and χ2 or Fisher's exact test, for categorical variables, will be used to summarize the data and compare characteristics between the 2 groups. The incidence of delirium will be compared using χ2 test and multivariable logistic regression. Differences in the duration of delirium and MV between the intervention and control groups will be analyzed by analysis of variance (ANOVA). The length of stay will be compared by truncated negative binomial regression, while mortality rates will be compared via logistic regression. A sensitivity analysis will be performed in order to assess the possible confounding effect of the non-randomized nature of our study design. A propensity score model for receipt of standard care vs. psychiatric involvement will be performed in order to approximate a balanced covariate distribution between the 2 groups as that would be expected by randomization. The investigators will then use the propensity score for each subject to perform an inverse probability weighted comparison of the groups on our trial outcomes.

ELIGIBILITY:
Inclusion criteria are:

1. Patients who are ≥18 years of age
2. Patients admitted to the surgical ICU for >48 hours OR
3. Patients admitted to the ICU <24 hours who have been in the hospital >48 hours

   OR
4. Patients who return to the ICU after being discharged from the ICU to the floor due a complication or need for higher acuity care.
5. Patients admitted to any surgical service who are receiving care in the 7 West surgical ICU, who are either medically or conservatively managed (non-surgical) or surgically managed as part of their care

Exclusion criteria are:

1. Patients in whom CAM-ICU cannot be performed (severe dementia, stroke or other neurological condition, encephalopathy, mental retardation, severe psychiatric disorder, vegetative state, severe traumatic brain injury, deaf/blind, etc.)
2. Patients who don't speak or understand English
3. Current alcohol or substance abuse
4. Patients who already have delirium within 24-48 hours of their ICU admission [Defined as a positive CAM-ICU test, or based on the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition ( DSM-V) diagnostic criteria:

   * Disturbance in attention (ie, reduced ability to direct, focus, sustain, and shift attention) and awareness.
   * Change in cognition (eg, memory deficit, disorientation, language disturbance, perceptual disturbance) that is not better accounted for by a preexisting, established, or evolving dementia.
   * The disturbance develops over a short period (usually hours to days) and tends to fluctuate during the course of the day.
   * There is evidence from the history, physical examination, or laboratory findings that the disturbance is caused by a direct physiologic consequence of a general medical condition, an intoxicating substance, medication use, or more than one cause.]

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Incidence of ICU delirium. | Average of one year.
  primary outcome measure is the incidence of ICU delirium.

SECONDARY OUTCOMES:
Duration of delirium. | Average of one year.
  Total days of delirium (even if they are non-consecutive).
Hospital length of stay | Average of one year.
  Total days of hospital length of stay.
Total days of mechanical ventilation. | Average of one year.
  In days.
In-hospital mortality | Average of one year.
  In-hospital mortality
ICU length of stay | Average of one year.
  Total days of ICU length of stay.

OTHER OUTCOMES:
Age | Average of one year.
  in years
Gender | Average of one year.
  male or female
Body mass index (BMI) | Average of one year.
  weight and height will be used to calculate BMI in kg/m^2
History of alcohol or substance abuse | Average of one year.
  any remote history; patients must be sober 6 months prior to study enrollment
Admitting diagnosis | Average of one year.
  Verbal admitting diagnosis (not using ICD codes)
Dementia | Average of one year.
  yes or no
Comorbid conditions | Average of one year.
  verbal list of other medical conditions
admitting Sequential Organ Failure Assessment (SOFA) score | Average of one year.
  Use MDCalc to calculate score using: admitting PaO2 (mmHg), FiO2 (%), platelets (x10^3/mcL), glasgow coma scale (points 3-15), bilirubin (mg/dL), level of hypotension (0-4 point scale based on mean arterial pressure value in mmHg, and the number and doses of vasopressors the patient is on), Creatinine (point assigned from 0-4 based on creatinine values ranging from Cr<1.2 mg/dL to Cr>5mg/dL)
Use of deliriogenic medications | Average of one year.
  List of medications which are known to be deliriogenic as described in literature and the 2018 American Geriatric Society Beers criteria which are administered to the participant.
Treatment of delirium | Average of one year.
  Description of intervention used to treat delirium (i.e. non pharmacological measures like family involvement) or medications (i.e. haloperidol). It will also be specified if the treatment was initiated by the ICU or psychiatry team.
Number of days from hospital admission to study enrollment | Average of one year.
  In days
height | Average of one year.
  measured in meters-used for BMI calculation
weight | Average of one year.
  Measured in kilograms (kg)-used for BMI calculation.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine M Kuza, MD, Principal Investigator — University of Southern California
Locations (1):
- Keck School of Medicine of the University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jackson P, Khan A. Delirium in critically ill patients. Crit Care Clin. 2015 Jul;31(3):589-603. doi: 10.1016/j.ccc.2015.03.011. Epub 2015 May 4. PMID 26118922
- [Result] Fong TG, Tulebaev SR, Inouye SK. Delirium in elderly adults: diagnosis, prevention and treatment. Nat Rev Neurol. 2009 Apr;5(4):210-20. doi: 10.1038/nrneurol.2009.24. PMID 19347026
- [Result] Brummel NE, Girard TD. Preventing delirium in the intensive care unit. Crit Care Clin. 2013 Jan;29(1):51-65. doi: 10.1016/j.ccc.2012.10.007. PMID 23182527
- [Result] Ely EW, Shintani A, Truman B, Speroff T, Gordon SM, Harrell FE Jr, Inouye SK, Bernard GR, Dittus RS. Delirium as a predictor of mortality in mechanically ventilated patients in the intensive care unit. JAMA. 2004 Apr 14;291(14):1753-62. doi: 10.1001/jama.291.14.1753. PMID 15082703
- [Result] van Eijk MM, van Marum RJ, Klijn IA, de Wit N, Kesecioglu J, Slooter AJ. Comparison of delirium assessment tools in a mixed intensive care unit. Crit Care Med. 2009 Jun;37(6):1881-5. doi: 10.1097/CCM.0b013e3181a00118. PMID 19384206
- [Result] Barr J, Fraser GL, Puntillo K, Ely EW, Gelinas C, Dasta JF, Davidson JE, Devlin JW, Kress JP, Joffe AM, Coursin DB, Herr DL, Tung A, Robinson BR, Fontaine DK, Ramsay MA, Riker RR, Sessler CN, Pun B, Skrobik Y, Jaeschke R; American College of Critical Care Medicine. Clinical practice guidelines for the management of pain, agitation, and delirium in adult patients in the intensive care unit. Crit Care Med. 2013 Jan;41(1):263-306. doi: 10.1097/CCM.0b013e3182783b72. PMID 23269131
- [Result] Hayhurst CJ, Pandharipande PP, Hughes CG. Intensive Care Unit Delirium: A Review of Diagnosis, Prevention, and Treatment. Anesthesiology. 2016 Dec;125(6):1229-1241. doi: 10.1097/ALN.0000000000001378. PMID 27748656
- [Result] Salluh JI, Latronico N. Making advances in delirium research: coupling delirium outcomes research and data sharing. Intensive Care Med. 2015 Jul;41(7):1327-9. doi: 10.1007/s00134-015-3864-4. Epub 2015 Jun 3. No abstract available. PMID 26077062
- [Result] Zhang H, Lu Y, Liu M, Zou Z, Wang L, Xu FY, Shi XY. Strategies for prevention of postoperative delirium: a systematic review and meta-analysis of randomized trials. Crit Care. 2013 Mar 18;17(2):R47. doi: 10.1186/cc12566. PMID 23506796
- [Result] Ringdal GI, Ringdal K, Juliebo V, Wyller TB, Hjermstad MJ, Loge JH. Using the Mini-Mental State Examination to screen for delirium in elderly patients with hip fracture. Dement Geriatr Cogn Disord. 2011;32(6):394-400. doi: 10.1159/000335743. Epub 2012 Feb 1. PMID 22301509
- [Result] Roberts DJ, Goralski KB, Renton KW, Julien LC, Webber AM, Sleno L, Volmer DA, Hall RI. Effect of acute inflammatory brain injury on accumulation of morphine and morphine 3- and 6-glucuronide in the human brain. Crit Care Med. 2009 Oct;37(10):2767-74. doi: 10.1097/CCM.0b013e3181b755d5. PMID 19865006
- [Result] Collinsworth AW, Priest EL, Campbell CR, Vasilevskis EE, Masica AL. A Review of Multifaceted Care Approaches for the Prevention and Mitigation of Delirium in Intensive Care Units. J Intensive Care Med. 2016 Feb;31(2):127-41. doi: 10.1177/0885066614553925. Epub 2014 Oct 27. PMID 25348864
- [Result] Kalabalik J, Brunetti L, El-Srougy R. Intensive care unit delirium: a review of the literature. J Pharm Pract. 2014 Apr;27(2):195-207. doi: 10.1177/0897190013513804. Epub 2013 Dec 10. PMID 24326408
- [Result] Slooter AJ, Van De Leur RR, Zaal IJ. Delirium in critically ill patients. Handb Clin Neurol. 2017;141:449-466. doi: 10.1016/B978-0-444-63599-0.00025-9. PMID 28190430
- [Result] Abelha FJ, Luis C, Veiga D, Parente D, Fernandes V, Santos P, Botelho M, Santos A, Santos C. Outcome and quality of life in patients with postoperative delirium during an ICU stay following major surgery. Crit Care. 2013 Oct 29;17(5):R257. doi: 10.1186/cc13084. PMID 24168808
- [Result] Van Rompaey B, Schuurmans MJ, Shortridge-Baggett LM, Truijen S, Elseviers M, Bossaert L. Long term outcome after delirium in the intensive care unit. J Clin Nurs. 2009 Dec;18(23):3349-57. doi: 10.1111/j.1365-2702.2009.02933.x. Epub 2009 Sep 4. PMID 19735334
- [Result] Pisani MA, Kong SY, Kasl SV, Murphy TE, Araujo KL, Van Ness PH. Days of delirium are associated with 1-year mortality in an older intensive care unit population. Am J Respir Crit Care Med. 2009 Dec 1;180(11):1092-7. doi: 10.1164/rccm.200904-0537OC. Epub 2009 Sep 10. PMID 19745202
- [Result] Turnbull AE, Neufeld KJ, Needham DM. Contradictory findings on one-year mortality following ICU delirium. Crit Care. 2015 Jan 30;19(1):29. doi: 10.1186/s13054-015-0747-6. No abstract available. PMID 25887540
- [Result] Leslie DL, Inouye SK. The importance of delirium: economic and societal costs. J Am Geriatr Soc. 2011 Nov;59 Suppl 2(Suppl 2):S241-3. doi: 10.1111/j.1532-5415.2011.03671.x. PMID 22091567
- [Result] van den Boogaard M, Schoonhoven L, Evers AW, van der Hoeven JG, van Achterberg T, Pickkers P. Delirium in critically ill patients: impact on long-term health-related quality of life and cognitive functioning. Crit Care Med. 2012 Jan;40(1):112-8. doi: 10.1097/CCM.0b013e31822e9fc9. PMID 21926597
- [Result] Davydow DS. Symptoms of depression and anxiety after delirium. Psychosomatics. 2009 Jul-Aug;50(4):309-16. doi: 10.1176/appi.psy.50.4.309. PMID 19687169
- [Result] Pandharipande PP, Girard TD, Jackson JC, Morandi A, Thompson JL, Pun BT, Brummel NE, Hughes CG, Vasilevskis EE, Shintani AK, Moons KG, Geevarghese SK, Canonico A, Hopkins RO, Bernard GR, Dittus RS, Ely EW; BRAIN-ICU Study Investigators. Long-term cognitive impairment after critical illness. N Engl J Med. 2013 Oct 3;369(14):1306-16. doi: 10.1056/NEJMoa1301372. PMID 24088092
- [Result] Marra A, Ely EW, Pandharipande PP, Patel MB. The ABCDEF Bundle in Critical Care. Crit Care Clin. 2017 Apr;33(2):225-243. doi: 10.1016/j.ccc.2016.12.005. PMID 28284292
- [Result] Holmes A, Hodgins G, Adey S, Menzel S, Danne P, Kossmann T, Judd F. Trial of interpersonal counselling after major physical trauma. Aust N Z J Psychiatry. 2007 Nov;41(11):926-33. doi: 10.1080/00048670701634945. PMID 17924246
- [Result] Rymaszewska J, Kiejna A, Hadrys T. Depression and anxiety in coronary artery bypass grafting patients. Eur Psychiatry. 2003 Jun;18(4):155-60. doi: 10.1016/s0924-9338(03)00052-x. PMID 12814847
- [Result] Khan BA, Lasiter S, Boustani MA. CE: critical care recovery center: an innovative collaborative care model for ICU survivors. Am J Nurs. 2015 Mar;115(3):24-31; quiz 34, 46. doi: 10.1097/01.NAJ.0000461807.42226.3e. PMID 25674682
- [Result] Desan PH, Zimbrean PC, Weinstein AJ, Bozzo JE, Sledge WH. Proactive psychiatric consultation services reduce length of stay for admissions to an inpatient medical team. Psychosomatics. 2011 Nov-Dec;52(6):513-20. doi: 10.1016/j.psym.2011.06.002. PMID 22054620
- [Result] Angel C, Brooks K, Fourie J. Standardizing Management of Adults with Delirium Hospitalized on Medical-Surgical Units. Perm J. 2016 Fall;20(4):16-002. doi: 10.7812/TPP/16-002. Epub 2016 Sep 9. PMID 27644045
- [Result] Peris A, Bonizzoli M, Iozzelli D, Migliaccio ML, Zagli G, Bacchereti A, Debolini M, Vannini E, Solaro M, Balzi I, Bendoni E, Bacchi I, Trevisan M, Giovannini V, Belloni L. Early intra-intensive care unit psychological intervention promotes recovery from post traumatic stress disorders, anxiety and depression symptoms in critically ill patients. Crit Care. 2011;15(1):R41. doi: 10.1186/cc10003. Epub 2011 Jan 27. PMID 21272307
- [Result] Papathanassoglou ED. Psychological support and outcomes for ICU patients. Nurs Crit Care. 2010 May-Jun;15(3):118-28. doi: 10.1111/j.1478-5153.2009.00383.x. PMID 20500650
- [Result] Beach SR, Chen DT, Huffman JC. Educational impact of a psychiatric liaison in the medical intensive care unit: effects on attitudes and beliefs of trainees and nurses regarding delirium. Prim Care Companion CNS Disord. 2013;15(3):PCC.12m01499. doi: 10.4088/PCC.12m01499. Epub 2013 Jun 6. PMID 24171148
- See also: Guastelli LR et al. Integral patient care: mental health in a critical patient service — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3124197/

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-03-20): https://cdn.clinicaltrials.gov/large-docs/95/NCT03550495/Prot_SAP_000.pdf
  • Informed Consent Form (2018-03-20): https://cdn.clinicaltrials.gov/large-docs/95/NCT03550495/ICF_001.pdf